CLINICAL TRIAL: NCT03249389
Title: Study Assessing the Changes in Markers of Calcium Vitamin Metabolism of Patients Taken in Charge by Chemotherapy for Breast Cancer Adjuvant
Brief Title: Assessing the Changes in Markers of Calcium Vitamin Metabolism of for Breast Cancer Adjuvant (CALCIOBS)
Acronym: CALCIOBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ICM-URC-2014/55
Record Dates: First submitted 2016-08-29; First posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2016-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood sample (Experimental): patients will have a blood sample of 20 ml (4 x 5ml) for inclusion, the J1 of each course and at the end of treatment
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — patients will have a blood sample of 20 ml (4 x 5ml) for inclusion, the J1 of each course and at the end of treatment

SUMMARY:
This study is to Assess hypercalciuria between J1 of the cure and 1 J1 6 of the cure of adjuvant chemotherapy in patients receiving conventional adjuvant chemotherapy of breast cancer.

DETAILED DESCRIPTION:
In view of the absence of data published on the changes of the vitamin and calcium metabolism in patients of a breast cancer receiving adjuvant chemotherapy combined with corticosteroids in antiemetic aiming and a basal calcium vitamin deficiency. A non randomized study evaluating the percentage of change in the vitamin and calcium balance and the occurrence of a hypercalciuria between initiation and the end of the adjuvant chemotherapy seems necessary, both from the scientific point of view, but also to estimate the usefulness of these markers in clinical practice track.

This study is to Assess hypercalciuria between J1 of the cure and 1 J1 6 of the cure of adjuvant chemotherapy in patients receiving conventional adjuvant chemotherapy of breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Mammary adenocarcinoma to receive 6 cycles of adjuvant chemotherapy.

  * Performance index according to who less than or equal to 1.
  * Patient older than 18 years and older.
  * Patient affiliated to a social security scheme or beneficiary of an equivalent French social protection system
  * The informed consent signed and before any procedures specific to the test screening.

    * Pregnancy test negative for women and a means of contraception for women and men of reproductive age

Exclusion Criteria:

* The presence of metastatic disease.

  * Other cancer (except basal-cell skin carcinoma and cancer of the cervix in situ treated adequately and curative) treated in the 3 previous years.
  * Contraindications for the calcium and colecalciferol:-severe hypersensitivity to vitamin D or calcium supplementation or any of the excipients
* Pathology and/or conditions causing a hypercalcemia and/or hypercalciuria
* Calcium lithiasis - tissue calcification
* Hypervitaminosis D • Presence of significant co-morbidities: Uncontrolled endocrine disease. Known disorders of the phospho-calcium balance in the last 3 years. Osteopenia or osteoporosis proven treatment vitamin and calcium.

  * Concomitant treatment with experimental products.
  * Pregnant or nursing
  * Legal incapacity or limited legal capacity. Medical or psychological conditions, allowing the subject to complete the study or to sign the consent (art.) L.1121 - 6, L.1121 - 7, L.1211 - 8, L1211-9).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Assess the percentage of occurrence of a hypercalciuria | through study completion, an average of 1 year
  Assess the percentage of occurrence of a hypercalciuria between the J1 of the cure 1 and day 1 of the 6 of the adjuvant chemotherapy treatment

SECONDARY OUTCOMES:
Assess of vitamin and calcium balance | through study completion, an average of 1 year
  evolution of the different biological markers of vitamin and calcium balance

CONTACTS AND LOCATIONS:
Overall Officials: William JACOT, Study Chair — Institut régional du Cancer de Montpellier
Locations (1):
- Institut régional du Cancer de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No